CLINICAL TRIAL: NCT05960279
Title: Microwave Imaging in NeuroTrauma (MINT) - a Feasibility Study Investigating Whether Microwave-based Scanning Technology Can Detect an Intra-cranial Bleed in Adult Head Injury Patients
Brief Title: Microwave Imaging in NeuroTrauma
Acronym: MINT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Air Ambulance Charity Kent, Surrey, Sussex (Unknown); St George's University Hospitals NHS Foundation Trust (Other); Medfield Diagnostics AB (Unknown)
Responsible Party: Sponsor
Other Study IDs: 223018
Record Dates: First submitted 2023-07-12; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Craniocerebral Trauma
Keywords: Head injury; Traumatic brain injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training group: The head CT findings from this patient group will be used to teach the MD100 how to interpret its scan of the patients.
  Interventions: Device: MD100
- Testing group: Once sufficient training data has been obtained, subsequent head CT findings from patients enrolled into the study will be used to test the accuracy of the MD100
  Interventions: Device: MD100

INTERVENTIONS:
Device: MD100 — The MD100 (Medfield Diagnostics, Gothenburg, Sweden) consists of 8 antennas and measurement electronics integrated into a single device; rechargeable ion batteries power the instrument. The radiation transmitted from the device equals approximately 1% of the radiation emitted from a mobile phone. The device is non-invasive and small enough that it can be moved around with ease.
  The system transmits microwaves with an output of 0.2 milliWatts (mW) for less than 90 seconds. The power absorbed by the body is 100mW/kg which is a factor of 200 less than what is established by the existing safety standard for microwaves. A mobile phone output, by comparison, can be up to 250mW.
  The patient's head is placed in the instrument during measurement while the patient is supine. The procedure takes, on average, 5 minutes to perform.

SUMMARY:
The study aims to investigate whether microwave-based technology can be used as a bedside decision-making aid to identify patients who may have a bleed in their head.

The MD100 is a microwave-based head scanner, developed for the purpose of detecting strokes. In clinical trials, it was noticed that the device performed better when the patient suffered a stroke due to a bleed. It was believed that this device had wider applications in trauma care.

The MD100 has demonstrated a very high level of accuracy in detecting bleeds in small clinical trials in the non-acute setting. The device is supported by software that determines the presence of a bleed.

This study will be set in the emergency department of major trauma centres. Patients that have sustained a head injury will be considered for enrollment into the study. Following a head CT scan, patients will be scanned by the MD100. The trial will run in two phases.

In phase one: the findings from the patient's head CT scan will be used to trial the device and teach the software what it is scanning. In phase two: The MD100 will be tested to see whether it can concur with the findings of the patient's CT scan, this will be used to determine the accuracy and reliability of the device.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and over.
* Blunt head trauma
* The patient has had a CT head scan

Exclusion Criteria:

* Patients with head injuries penetrating the skull
* Patients with radiologically confirmed cervical spine fracture
* Patients with radiologically confirmed depressed skull fracture and/or dislocation
* Patients with implanted metal in or around their skull (including titanium places and surgical staples)
* Confirmed pregnancy
* Per the investigator's judgement, any condition or symptoms preventing the patient from entering the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head injury patients presenting to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the MD100 | One year
  The MD100's proportion of true positives of intracranial bleeds detected in the head injured patient.

CONTACTS AND LOCATIONS:
Overall Officials: Malcom Tunnicliff, MBBS, Study Director — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - King's College Hospital NHS FT, London
  - St George's Hospital NHS FT, London

IPD SHARING:
Plan to Share IPD: Undecided